CLINICAL TRIAL: NCT01817842
Title: Comparative Effectiveness of Web-based Mobile Support for the DC Tobacco Quitline
Brief Title: Study of Mobile Phone Support for the DC Tobacco Quitline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Truth Initiative (Other)
Responsible Party: Principal Investigator, Thomas Kirchner, Research Investigator, Truth Initiative
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC1DA028710 (NIH)
Record Dates: First submitted 2013-03-20; First posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Smoking Cessation
Keywords: mHealth; EMA; Ecological Momentary Assessment; Personal Informatics; Tobacco Quitline
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mEX support (Experimental): Participants in this arm receive both standard DC Quitline Support and Mobile EX cessation support. Mobile EX cessation support is designed to enhance the Washington D.C. Quitline (DCQL) by giving participants the ability track their cessation attempt on a phone-based app and thus create a profile documenting their progress and set-backs over the days or weeks in between QL contacts. Participants receive summary information and graphics that help them understand what is working best for them. Participants also receive 24-hr, momentary access to a set of interactive cessation tools on their phone.
  Interventions: Behavioral: Mobile EX cessation support; Behavioral: DC Quitline Support
- Device Control (Active Comparator): Participants randomized to this arm receive standard DC Quitline Support plus the device control. Device control includes an identical device (i.e., mobile phone) to that provided to the intervention group, but participants do not receive any of the phone-based mEX support features. Those in the device control group receive their device at the 1-month time point - a design feature that allows a direct comparison of the mEX intervention to standard quitline services over the first month.
  Interventions: Behavioral: DC Quitline Support; Behavioral: Device Control

INTERVENTIONS:
Behavioral: Mobile EX cessation support — Mobile EX cessation support is designed to enhance the Washington D.C. Quitline (DCQL) by giving participants the ability track their cessation attempt on a phone-based app and thus create a profile documenting their progress and set-backs over the days or weeks in between QL contacts. Participants receive summary information and graphics that help them understand what is working best for them. Participants also receive 24-hr, momentary access to a set of interactive cessation tools on their phone.
  Other Names: mEX
  Arms: mEX support
Behavioral: DC Quitline Support — Participants assigned to standard DC Quitline programming receive 6 proactive QL counseling sessions and optional, free nicotine replacement therapy (NRT).
Behavioral: Device Control — Mobile phone for use during cessation attempt but with no mEX support components
  Arms: Device Control

SUMMARY:
This is a study of the effectiveness of mobile phone support for the D.C. Tobacco Quitline. The project will test the efficacy of a web-based system that uses mobile phones to improve quit rates at 3-month intervals, relative to standard quitline services. Under the standard model, relatively infrequent, periodic support is provided to smokers who want to quit and seek out the services. The new system will complement that effort by increasing the quality, frequency and accessibility of quit smoking support - when and where the smoker needs it most. It is hypothesized that successful abstinence rates will improve to the degree that participants utilize the support system and engage with the quitline.

DETAILED DESCRIPTION:
This study aims to bolster the effectiveness of the Washington D.C. Quitline (DCQL) program with the addition of a web-based mobile EX (mEX) cessation support system. This mEX system is designed to fill the gaps between quitline calls with ready access to a menu of evidenced-based treatment components, while also providing DCQL counselors with detailed information about their clients' ongoing progress with cessation - two developments that constitute a major advance over standard quitline programming. With the addition of mEX, DCQL counselors will be able to tailor their advice from the outset of each call and even identify counterproductive patterns that would have otherwise gone unnoticed. This innovative extension of our previous work leverages our expertise with ecological assessment methodology and behavioral informatics for the purpose of dynamic relapse prevention support within the context of an underserved community QL.

The project is an additive two-group randomized controlled trial to test whether the addition of mEX improves abstinence rates at 1-, 3-, 6-, and 9-months relative to standard care provided by DCQL. Participants will be 700 smokers who contact the DCQL and are randomized to receive either standard DCQL programming (N=300) or DCQL plus MQE (N=400). Participants assigned to standard DCQL programming will receive 6 proactive QL counseling sessions and free nicotine replacement therapy (NRT). Participants assigned to DCQL plus MQE will also receive mobile access to the MQE system via a web-enabled cellular telephone provided by the study. Relative to usual care, we expect that MQE will improve outcomes by improving delivery, utilization and thereby effectiveness of DCQL resources.

Specific Aim 1. Examine abstinence rates in DCQL participants receiving usual-care relative to those also receiving mobile quitline enhancement. Relative to usual-care controls, mobile quitline enhancement is expected to improve 7-day point prevalence abstinence rates at 1-, 3-, 6-, and 9-months.

Specific Aim 2. Examine treatment utilization in DCQL participants receiving usual-care relative to those also receiving mobile quitline enhancement. Relative to usual-care controls, mobile quitline enhancement is expected to improve utilization of available DCQL programming resources.

Specific Aim 3. Examine whether utilization of DCQL or mobile support services moderates their impact on outcomes. Treatment effects are expected to vary with the degree that they are utilized, such that greater utilization will predict improved abstinence rates at all time points.

ELIGIBILITY:
Inclusion Criteria:

* Active tobacco smoker of at least 5 cigarettes / day
* Read, speak and write English
* Access to a telephone at either home or work
* Contacts DC Tobacco Quitline and makes an attempt to quit smoking

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Smoking Abstinence | 9-months
  Point-prevalent abstinence from smoking cigarettes over the past 7-days. Verified with expired carbon monoxide at 1-month. Reported by participants at 3-, 6- and 9-months.

SECONDARY OUTCOMES:
Daily Lapse Status | Month 1
  Daily abstinence versus any smoking (i.e., lapse) status among those who are actively trying to abstain (i.e., not those who have completely relapsed).
Quitline utilization | Month 1
  Participant receipt and initiation of support calls from DC Quitline staff.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kirchner, PhD, Principal Investigator — Truth Initiative
Locations (1):
- United Medical Center, Washington D.C., District of Columbia, United States